CLINICAL TRIAL: NCT03442686
Title: Compass Course: Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CKMW-1801
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a wait list control design. One group of participants will be evaluated before receiving the intervention (in Spring 2018) and compared to those who receive the intervention in Spring 2018. The first group will go on to receive the intervention in Fall 2018.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spring 2018 Compass Course Group (Experimental): Two groups of up to 15 participants (30 total) will receive the study intervention during Spring 2018. All participants will complete study questionnaires before and after the Spring sessions.
  Interventions: Behavioral: Compass Course
- Spring 2018 Comparison Group (No Intervention): Two groups of up to 15 participants will receive the study intervention in Fall 2018. All participants will complete study questionnaires before and after the Spring sessions. Those who enroll in the study and agree to participate in the Fall sessions will serve as a no-treatment comparison group.

INTERVENTIONS:
Behavioral: Compass Course — An 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention, called the Compass Course is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in their daily lives.
  Arms: Spring 2018 Compass Course Group

SUMMARY:
The Compass Course is an 8-session progressive structure that was developed based on theoretical and scientific evidence from psychology and occupational therapy. The goal of the intervention is to provide participants with information, tools, and support that help them move towards reclaiming a sense of self-grounded purpose in daily life. The study will use a convenience sample of breast cancer survivors to evaluate the efficacy of the Compass Course intervention.

ELIGIBILITY:
Inclusion criteria:

1. 25 years of age or older
2. Completed treatment (such as chemotherapy, radiation, surgery) for Stage 0, 1, 2, or 3 breast cancer at least 2 months prior to participating in the Compass Course intervention
3. English speaking
4. High school diploma or GED
5. Able to see, hear, speak (with or without assistive devices)
6. Able to provide own transportation to sessions
7. Willing and able to commit to attend all 8 intervention sessions

Exclusion criteria (all self-reported):

1. Stage 4 breast cancer or any other stage 4 cancer
2. Actively receiving chemotherapy or radiation treatments for cancer. (However, patients may be on Herceptin and/or endocrine treatment and participate in the study.)
3. History of neurologic disorder (such as stroke or brain injury) with residual impairments that likely interfere with learning
4. Any medical condition (physical or mental health) that interferes with the performance of everyday activities and roles.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in psychological well-being | Will be administered at Week 0 (pre-testing), at Week 12 (session 8), and at 3 month follow up
  Using the Psychological Scales of Wellbeing questionnaire (Ryff, 1989; Ryff, & Keyes, 1995), psychological wellbeing pre- and post- intervention will be tracked.

SECONDARY OUTCOMES:
Recruitment | Up to 1 month after IRB approval
  Number of prospective participants approached by clinicians and number of self-referred prospective participants who contact PI or Study Coordinator with inquiries about the study
Time of pre-testing session | Duration of pre-testing session (approximately 2 hours) at week 0 to week 1
  Actual length (in minutes) of pre-testing session.
Time of testing session | Each week from week 2 through week 8, approximately 2 hours at each session
  Actual length (in minutes) of testing session.
Time of post-testing session | Duration of session 8 (at week 12), approximately 1 hour
  Actual length (in minutes) of testing session.
Homework completion | Each week from week 2 through week 8
  Whether or not homework was attempted
Intervention fidelity | Each week from week 2 through week 8
  Which key intervention elements were provided during a given session
Change in Meaning in life | At week 0 and at week 12, and at 3 month follow up
  Meaning in Life Questionnaire (Steger et al., 2006): A 10-item questionnaire designed to measure 2 dimensions of meaning in life: Presence of Meaning (how much respondents feel their lives have meaning) and Search for Meaning (how much respondents strive to find meaning and understanding in their lives).
Engagement in Meaningful Activities | At week 0 and at week 12
  Engagement in Meaningful Activities Survey (Eakman, 2010):A 12-item self-report questionnaire designed to measure the extent to which a person experiences meaningfulness in his/her daily life activities.
Purpose Status and Expectations | At week 0, at week 12, and at 3 month follow up
  A 2-question self-report developed by the study team to better understand what participants' hope to gain during the study and perceived changes.
Participant Experience of Compass Course | At week 12 and at week 14-20
  Participant experience of Compass Course as measured by self-report questionnaire and post-intervention focus group.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Radomski, PhD, OTR/L, Principal Investigator — Allina Health
Locations (3):
- United States (3):
  - Courage Kenny Rehabilitation Institute, Golden Valley, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Shoreview Clinic, Shoreview, Minnesota